CLINICAL TRIAL: NCT03934216
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Efficacy of BMS-986165 in Subjects With Moderate to Severe Ulcerative Colitis
Brief Title: Safety and Efficacy of Deucravacitinib in Participants With Moderate to Severe Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-024; 2018-004694-27 (EudraCT Number)
Record Dates: First submitted 2019-04-30; First posted 2019-05-01 (Actual); Results first posted 2022-07-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-02

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BMS-986165 (Experimental)
  Interventions: Drug: BMS-986165
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified Dose on Specified Days
  Other Names: Deucravacitinib
  Arms: BMS-986165
Other: Placebo — Specified Dose on Specified Days
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and efficacy of oral deucravacitinib in participants with moderate to severe ulcerative colitis (UC).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Must have active ulcerative colitis (UC) extending ≥ 15 cm from the anal verge and confirmed by a screening/baseline colonoscopy/sigmoidoscopy prior to the randomization visit
* Must have documented diagnosis of UC of at least 3 months' duration prior to screening
* Must have active moderate to severe UC, as defined by a modified Mayo score of 5 to 9 points, inclusive, which includes a stool frequency (SF) subscore of ≥ 2, and a rectal bleeding (RB) subscore ≥ 1, and a screening endoscopic (ES) subscore of ≥ 2

Exclusion Criteria:

* Previous/current documented diagnosis of CD, indeterminate colitis, ischemic colitis, or pseudomembranous colitis (other than associated with Clostridium difficile [C. difficile])
* Stool positive for C. difficile toxin at screening visit
* Current or recent (within 12 weeks prior to the randomization visit) evidence of fulminant colitis, abdominal abscess, toxic megacolon, or bowel perforation

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-13 (Actual); Study Completion 2023-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (104):
- United States (30):
  - Connecticut Clinical Research Foundation, Bristol, Connecticut
  - University of Florida, Gainesville, Florida
  - Local Institution - 0048, New Port Richey, Florida
  - Local Institution - 0044, Sweetwater, Florida
  - Local Institution - 0011, Suwanee, Georgia
  - Local Institution - 0121, Glenview, Illinois
  - Texas Digestive Disease Consultants - Gastroenterology Associates - Baton Rouge, Baton Rouge, Louisiana
  - Local Institution - 0018, Shreveport, Louisiana
  - Local Institution - 0047, Chevy Chase, Maryland
  - Infusion Associates, Grand Rapids, Michigan
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Local Institution - 0002, Las Vegas, Nevada
  - Local Institution - 0049, Lake Success, New York
  - New York University Langone Medical Center, New York, New York
  - Consultants for Clinical Research, Cincinnati, Ohio
  - Penn State Health Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Local Institution - 0074, Charleston, South Carolina
  - Rapid City Medical Center, Rapid City, South Dakota
  - Gastro One, Germantown, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Local Institution - 0097, Garland, Texas
  - Local Institution - 0008, Houston, Texas
  - Gastroenterology Research of San Antonio, San Antonio, Texas
  - Local Institution - 0106, San Antonio, Texas
  - Texas Digestive Disease Consultants - Southlake, Southlake, Texas
  - Local Institution - 0116, Tyler, Texas
  - Local Institution - 0096, Seattle, Washington
  - Swedish First Hill Campus, Seattle, Washington
  - Local Institution - 0122, Vancouver, Washington
- Australia (4):
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Local Institution - 0071, Bedford Park, South Australia
  - Local Institution - 0108, Melbourne, Victoria
  - Fiona Stanley Hospital, Murdoch, Western Australia
- Belgium (3):
  - Local Institution - 0039, Antwerp
  - Local Institution - 0065, Brussels
  - Clinique du MontLegia - CHC, Liège
- Czechia (2):
  - Hepato-Gastroenterology HK, Hradec Králové
  - Nemocnice Slany, Slaný
- France (4):
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - Centre Hospitalier Universitaire de Saint-Etienne - Hopital Nord, Saint-Etienne
  - Local Institution, Toulouse
- Germany (6):
  - Charite Universitatsmedizin Berlin - Campus Virchow-Klinikum, Berlin
  - Universitatsklinikum Carl Gustav Carus Dresden, Dresden
  - Medizinische Hochschule Hannover, Hanover
  - Local Institution - 0070, Kiel
  - Local Institution - 0062, Leipzig
  - Universitatsklinik Ulm, Ulm
- Hungary (5):
  - Magyar Honvedseg-Egeszsegugyi Kozpont, Budapest
  - Local Institution - 0042, Budapest
  - Local Institution - 0024, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Bugat Pal Korhaz, Gyöngyös
- Italy (9):
  - Local Institution - 0033, Rozzano, Milano
  - Azienda Ospedaliero-Universitaria di Bologna - Policlinico SantOrsola-Malpighi, Bologna
  - Local Institution - 0005, Catanzaro
  - Clinica Medica Azienda Ospedaliera Universitaria, Messina
  - Azienda Ospedaliera di Padova, Padua
  - Local Institution - 0027, Pavia
  - Policlinico Universitario Campus Bio-Medico, Roma
  - Local Institution - 0046, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli, Roma
- Japan (10):
  - National Hospital Organization Hirosaki National Hospital, Hirosaki, Aomori
  - Fukuoka University Chikushi Hospital, Chikushino-shi, Fukuoka
  - Local Institution - 0078, Kurume, Fukuoka
  - National Hospital Organization Takasaki General Medical Center, Takasaki, Gunma
  - Hyogo College of Medicine Hospital, Nishinomiya, Hyōgo
  - Local Institution - 0081, Sagamihara-shi, Kanagawa
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Local Institution - 0066, Bunkyo-ku, Tokyo
  - Local Institution - 0080, Minato-ku, Tokyo
  - Local Institution - 0069, Saga
- Poland (16):
  - Local Institution - 0091, Bydgoszcz
  - Local Institution - 0013, Bydgoszcz
  - Local Institution - 0100, Lodz
  - Local Institution - 0045, Lodz
  - Local Institution - 0098, Nowy Targ
  - Local Institution - 0094, Piotrkow Trybunalski
  - Local Institution - 0040, Sopot
  - Local Institution - 0053, Szczecin
  - Local Institution - 0014, Tychy
  - Centrum Zdrowia Matki Dziecka i Mlodziezy, Warsaw
  - Local Institution - 0088, Warsaw
  - Local Institution - 0095, Warsaw
  - Niepubliczny Zaklad Opieki Zdrowotnej VIVAMED Jadwiga Miecz, Warsaw
  - Local Institution - 0030, Warsaw
  - Local Institution - 0037, Wroclaw
  - Centrum Medyczne Oporow, Wroclaw
- Russia (6):
  - Nizhniy Novgorod Regional Clinical Hospital N.A. Semashko, Nizhny Novgorod
  - Local Institution - 0020, Novosibirsk
  - Novosibirsk State Regional Clinical Hospital, Novosibirsk
  - Local Institution - 0092, Novosibirsk
  - Local Institution - 0015, Saratov
  - Multidisciplinary Consultative and Diagnostic Center, Tyumen
- South Korea (4):
  - Local Institution - 0064, Daegu
  - Local Institution, Daegu
  - Local Institution, Incheon
  - Local Institution, Seoul
- United Kingdom (5):
  - Barnsley Hospital NHS Foundation Trust, Barnsley
  - Local Institution - 0031, Cambridge
  - NHS Greater Glasgow and Clyde, Glasgow
  - Imperial College Healthcare NHS Trust, London
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/us/en/home.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 131 Participants Randomized and 129 Treated
Groups:
- Treatment: BMS-986-165 6mg BID
- Placebo: Placebo
Period: Overall Study
Arm/Group | Treatment | Placebo
Started | 88 | 43
Completed | 30 | 12
Not Completed | 58 | 31
Not completed — Other Reasons | 5 | 5
Not completed — Adverse Event | 22 | 11
Not completed — Lack of Efficacy | 8 | 7
Not completed — Lost to Follow-up | 2 | 0
Not completed — Non-Compliance with Study Drug | 1 | 1
Not completed — Pregnancy | 1 | 0
Not completed — Withdrawal by Subject | 18 | 6
Not completed — Randomized but not treated | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment | Placebo | Total
Number analyzed (Participants) | 88 | 43 | 131
Age, Continuous [Mean (Standard Deviation); unit: Years] | 41.6 (14.81) | 40.3 (13.91) | 41.2 (14.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 14 | 54
  Male | 48 | 29 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 83 | 41 | 124
  Unknown or Not Reported | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 7 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 80 | 34 | 114
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission Response Rate at Week 12
Description: Clinical remission response rate is the percentage of participants achieving clinical remission, defined as absolute total Mayo Score and absolute Mayo endoscopy, stool frequency, rectal bleeding.
  Will be calculated using a modified Mayo score with the following:
  Stool Frequency (SF) sub score ≤ 1, with ≥ 1 point decrease from baseline, and Rectal Bleeding (RB) sub score = 0, and Endoscopic (ES) sub score ≤ 1 (modified, excludes friability)
  The modified Mayo score (0 to 9 points) is the sum of 3 components: the SF, RB, and ES sub scores
  Modified Mayo Score: The modified Mayo score is a 9-point scale; a score of 5 to 9 points (inclusive), which is required for randomization, denotes moderate to severe disease (by protocol definition). considered in clinical remission if a Mayo Score of less than or equal to 2 with no individual sub score greater than 1
Time Frame: From first dose to 12 weeks.
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 88 | 43
Percentage of Participants | 14.8 [7.4 to 22.2] | 16.3 [5.2 to 27.3]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.5935, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.9, 95% CI 2-sided [0.3 to 2.4]

2. Secondary Outcome: Clinical Response Rate at 12 Weeks
Description: Clinical response is defined as percentage of participants with a reduction in total Mayo Score and reduction in rectal bleeding subscore
  Will be defined as the following:
  A decrease from baseline in the modified Mayo score of ≥ 2 points, and A decrease from baseline in the modified Mayo score ≥ 30%, and A decrease in rectal bleeding(RB) subscore of ≥ 1 point or absolute RB subscore ≤ 1
Time Frame: From first dose to 12 weeks
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 88 | 43
Percentage of participants | 37.5 [27.4 to 47.6] | 32.6 [18.6 to 46.6]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.3051, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.2, 95% CI 2-sided [0.6 to 2.7]

3. Secondary Outcome: Endoscopic Response at Week 12
Description: Endoscopic response will be defined as percentage of participants with a reduction in the total Ulcerative Colitis Endoscopic Index of Severity score.
  The Ulcerative Colitis Endoscopic Index of Severity (UCEIS) scale:
  Vascular Pattern:
  * Normal (score 0)
  * patchy obliteration (score 1)
  * Obliterated (score 2)
  Bleeding
  * None (score 0)
  * Mucosal (score 1)
  * Luminal mild (score 2)
  * Luminal Moderate or severe (score 3)
  Erosions and Ulcers
  * None (score 0)
  * Erosions ( score 1)
  * Superficial Ulcer (2)
  * Deep Ulcer (score 3)
  A total score represents the following: remission (0-1); mild (2-4); moderate (5-6); and severe (7-8).
Time Frame: up to 12 Weeks
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 88 | 43
Percentage of Participants | 19.3 [11.1 to 27.6] | 27.9 [14.5 to 41.3]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.8764, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 0.6, 95% CI 2-sided [0.3 to 1.4]

4. Secondary Outcome: Histological Improvement Response Rate at 12 Weeks
Description: Histologic improvement is defined as percentage of participants with a Geboes score of ≤ 3.1
  Neutrophils <5% of crypts, with no crypt destruction, erosions, ulcerations, and granulation tissue.
  Achieving the following scores for the corresponding grades of the Geboes score:
  * Score of 0 or 1 for Grade 3 (neutrophils in the epithelium: none or < 5% crypts involved), and
  * Score of 0 for Grade 4 (crypt destruction: none), and
  * Score of 0 Grade 5 (erosion or ulceration: no erosions, ulcerations, or granulation tissue)
  grade 1 = chronic inflammatory infiltrate; grade 2 = lamina propria neutrophils and eosinophils; grade 3 = neutrophils in the epithelium; grade 4 = crypt destruction; grade 5 = erosions or ulceration. A higher score indicates more severe disease
Time Frame: up to 12 Weeks
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Treatment | Placebo
Number analyzed (Participants) | 88 | 43
Percentage of Participants | 21.6 [13.0 to 30.2] | 16.3 [5.2 to 27.3]
Statistical Analysis 1: Comparison: Treatment vs Placebo; Test type: Superiority; p = 0.2235, Stratified Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.4, 95% CI 2-sided [0.5 to 3.8]

ADVERSE EVENTS:
Time Frame: Adverse Events and Serious Adverse Events: (From first dose to last dose + 100 days): Approximately 104 Weeks All-Cause mortality (From randomization to end of study): Approximately 104 Weeks
Description: The number at Risk for All-Cause Mortality represents all treated participants. The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication
Groups:
- BMS-986165 6mg BID During OL Period After Receiving Placebo in Induction Period: BMS-986165 6mg BID during OL period after receiving Placebo in Induction period
Arm/Group | Treatment | Placebo | BMS-986165 6mg BID During OL Period After Receiving Placebo in Induction Period
All-Cause Mortality (participants affected / at risk) | 2/87 | 0/10 | 0/32
Serious Adverse Events (participants affected / at risk) | 19/87 | 2/10 | 4/32
Other Adverse Events (participants affected / at risk) | 64/87 | 6/10 | 22/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=87) | Placebo (N=10) | BMS-986165 6mg BID During OL Period After Receiving Placebo in Induction Period (N=32)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Congenital aural fistula (Congenital, familial and genetic disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Colitis ulcerative (Gastrointestinal disorders) | 3 | 1 | 2
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 8 | 0 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
Nasal septum deviation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=87) | Placebo (N=10) | BMS-986165 6mg BID During OL Period After Receiving Placebo in Induction Period (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 7 | 0 | 1
Aphthous ulcer (Gastrointestinal disorders) | 5 | 1 | 2
Colitis ulcerative (Gastrointestinal disorders) | 17 | 2 | 8
Constipation (Gastrointestinal disorders) | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2
Fatigue (General disorders) | 1 | 0 | 2
Feeling cold (General disorders) | 0 | 0 | 2
Pyrexia (General disorders) | 3 | 0 | 5
Seasonal allergy (Immune system disorders) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 2
COVID-19 (Infections and infestations) | 13 | 0 | 6
Influenza (Infections and infestations) | 3 | 1 | 2
Nasopharyngitis (Infections and infestations) | 6 | 0 | 4
Oral herpes (Infections and infestations) | 2 | 1 | 1
Sinusitis (Infections and infestations) | 5 | 0 | 1
Tonsillitis (Infections and infestations) | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 5 | 0 | 1
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 1 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 2
Hepatitis B DNA assay positive (Investigations) | 0 | 1 | 0
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 0 | 4
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 9 | 0 | 2
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 13 | 0 | 3
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-14): https://cdn.clinicaltrials.gov/large-docs/16/NCT03934216/Prot_SAP_000.pdf